CLINICAL TRIAL: NCT00350961
Title: Phase I-II Study of bi-Weekly Fixed Dose Rate Gemcitabine, Oxaliplatin and Capecitabine in Patients With Advanced Cholangiocarcinoma
Brief Title: Gemcitabine, Oxaliplatin and Capecitabine in Patients With Advanced Cholangiocarcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Henrik Jensen, Dept. of Oncology, Vejle Sygehus, Vejle, Denmark (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEMOXEL cholangiocarcinoma
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Fixed dose rate; Gemcitabine; Oxaliplatin; Capecitabine
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine; Oxaliplatin; Capecitabine

INTERVENTIONS:
Drug: Gemcitabine
Drug: Oxaliplatin
Drug: Capecitabine

SUMMARY:
In Denmark approximately 200 new cases of cholangiocarcinoma are diagnosed every year. No standard treatment exists for patients with advanced cholangiocarcinoma, and improved systemic treatments are needed.

Duplets of gemcitabine, oxaliplatin and capecitabine have been evaluated in various cancers and several different regimens are well tolerated and active, especially in upper gastrointestinal cancers, exocrine pancreatic cancer and non-small cell lung cancer.

The triplet combination of these agents has not been studied, but a triplet combination of gemcitabine, oxaliplatin and 5-FU infusion has been evaluated in a phase I study.

Bi-weekly combination of gemcitabine and oxaliplatin has proven active and tolerable and warrants further study. In addition, fixed dose rate infusion of gemcitabine has shown interesting as the ability of mononuclear cells to accumulate gemcitabine triphosphate during therapy seems to be saturable.

We propose a phase I-II study of a bi-weekly schedule of gemcitabine, oxaliplatin and capecitabine. This regimen could be feasible in an out-patients setting.

The phase I part is a standard dose escalation study for patients with solid tumors. In the phase II part the recommended dose is studied in patients with advanced cholangiocarcinoma.

DETAILED DESCRIPTION:
Design

Open, non-randomized phase I/II study.

Purpose:

Phase I part To find MTD and RFTD for the combination of gemcitabine, oxaliplatin and capecitabine.

Dose Escalating Schedule Dose level Dose Gemcitabine 10 mg/m2/min 600-1000 mg/m2 day 1 and 14 Capecitabine p.o. x 2 daily. 1000-1250 mg/m2 day 1-7 and 14-21 Oxaliplatin 60-80 mg/m2day 1 and 14 Drugs: G C O Level 1 600 1000 60 Level 2 800 1000 60 Level 3 1000 1000 60 Level 4 1000 1250 60 Level 5 1000 1250 80 Level 6 1200 1250 80 Start level: Level 1, 3 patients per level

Phase II part The primary endpoint is the objective response rate The secondary endpoint is toxicity, response duration and time to progression.

Treatment:

Gemcitabine Gemcitabine is given intravenously on day 1 and 14 with a fixed dose rate of 10 mg/m2/min.

Oxaliplatin Oxaliplatin is given intravenously on day 1 and 14 as a 2 hours infusion.

Capecitabine Capecitabine is given orally and administered in tablets of 150 mg and 500 mg. The dose is administered twice daily with 12 hours interval, in the morning and evening during or latest 30 minutes after a meal.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven intra- or extrahepatic cholangiocarcinoma, papilla of the Vater or gallbladder carcinoma.
* PS 0-2
* Age 18-75
* Life expectancy > 12 weeks
* Normal bone marrow function (neutrophiles > 1,5 x 109/l and platelets > 100 x 109/l)
* Bilirubin < 1,5 x UNL
* Transaminases < 3 x UNL
* Normal renal function, Cr-EDTA clearance > 50 ml/min
* No chemotherapy, radiotherapy or immunotherapy 4 weeks prior to inclusion
* No known DPD-deficiency
* No neuropathy
* No uncontrolled, severe concurrent medical disease
* Signed informed consent

Exclusion Criteria:

* Chemotherapy, radiotherapy or immunotherapy 4 weeks prior to inclusion
* Experimental therapy < 8 weeks prior to inclusion
* Uncontrolled, severe concurrent medical disease
* Prior malignancy during the last 5 years, except for non-melanoma skin cancer and carcinoma in situ cervix uteri.
* Allergy to gemcitabine, oxaliplatin or capecitabine
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2004-06; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Response

SECONDARY OUTCOMES:
Safety
Time to progression
SUrvival

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Lassen, MD., PH.D., Principal Investigator — Rigshospitalet, Dept. of Oncology
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Vejle Sygehus, Vejle